CLINICAL TRIAL: NCT05708352
Title: A Randomized Controlled Phase 2 Study of the Ketogenic Diet Versus Standard Dietary Guidance for Patients With Newly Diagnosed Glioblastoma in Combination With Standard-of-care Treatment
Brief Title: A Phase 2 Study of the Ketogenic Diet vs Standard Anti-cancer Diet Guidance for Patients With Glioblastoma in Combination With Standard-of-care Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jethro Hu, Sponsor-Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022-06-HU-DIET2TREAT; R01CA276919 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
Keywords: Keto Diet
MeSH Terms: conditions — Glioblastoma | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keto-Diet (Experimental): Intensive 18-week Keto Diet intervention.
  Interventions: Behavioral: Keto Diet
- Standard Anti-Cancer Diet (Placebo Comparator): Standard Anti-Cancer Diet with Dietitian support
  Interventions: Behavioral: Standard Anti-Cancer Diet

INTERVENTIONS:
Behavioral: Keto Diet — The experimental intervention includes a strict and controlled diet that manages daily macronutrient breakdown and increases the ratio of dietary fat relative to protein and carbohydrate consumption.
  Arms: Keto-Diet
Behavioral: Standard Anti-Cancer Diet — Dietitian sessions will utilize the American Institute for Cancer Research Food resources and will reference foods low in fats such as fruits, vegetables and whole grains, providing key micronutrients and phytonutrients. Sessions will also focus on dietary support to help decrease any treatment related symptoms.
  Arms: Standard Anti-Cancer Diet

SUMMARY:
This is a Phase 2, randomized two-armed, multi-site study of 170 patients with newly diagnosed glioblastoma multiforme. Patients will be randomized 1:1 to receive Keto Diet, or Standard Anti-Cancer Diet. All patients will receive standard of care treatment for their glioblastoma. The Keto Diet intervention will be for an 18-week period and conducted by trained research dietitians. Daily ketone and glucose levels will be recorded to monitor Keto Diet adherence.

This two-armed randomized multi-site study aims to provide evidence to support the hypothesis that a Keto Diet vs. Standard Anti-Cancer Diet improves overall survival in newly diagnosed glioblastoma multiforme patients who receive standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Newly diagnosed glioblastoma (Within 2 months of initial diagnosis by histopathology)
* Not started standard of care chemotherapy and/or radiation therapy for glioblastoma
* Karnofsky Performance Status (KPS) ≥ 70
* Ability to read, write and understand either English OR Spanish
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Patients with recurrent glioblastoma
* Genetic disorders that affect lipid metabolism. Including but not limited to pyruvate carboxylase deficiency, porphyria, primary carnitine deficiency, carnitine palmitoyltransferase I or II deficiency, carnitine translocase deficiency, beta-oxidation defects
* Inability to wean steroids below 8mg dexamethasone / day or equivalent
* Body Mass Index (BMI) < 21kg/m2, unless the site Principal Investigator deems safe
* Currently pregnant or nursing
* Patients receiving other experimental therapy Note: Off-label therapy use is permitted
* Comorbidities that in the opinion of the investigator limit the patient's ability to complete the study
* Food preferences incompatible with keto diet
* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, cochlear implants (removable hearing aids permitted), or other electronic medical equipment, unless the site Principal Investigator deems safe
* Inability to participant in standard of care MRIs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From Baseline to 18 Months
  Will be calculated as the number of days from the date of patient registration to the date of death.

SECONDARY OUTCOMES:
Health-related quality of life 1 | From Baseline to 18 Weeks
  Measured by changes in the Functional Assessment of Cancer Therapy - Brain (FACT-BR) survey scores. Scores can range from 0- 200, the higher the score the better the quality of life.
Health-related quality of life 2 | From Baseline to 18 Weeks
  Measured by changes in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) survey scores. Scores can range from 0- 160, the higher the score the better the quality of life.
Progression-free survival | From Baseline to 18 Weeks
  Assessed with Magnetic resonance imaging (MRI) scan of the brain with and without gadolinium. MRI's will be reviewed and assessed for progression free survival via the modified Response Assessment in Neuro-Oncology Criteria.
Cognitive performance 1 | From Baseline to 18 Weeks
  Measured by changes in the Hopkins Verbal Test (HVLT-R) survey scores. Scores can range from 0-36, higher the scores the better the cognitive performance.
Cognitive performance 2 | From Baseline to 18 Weeks
  Measured by changes in the Trail Marking Test A/B survey scores. The longer the task takes to complete the lower the cognitive performance.
Physical activity | From Baseline to 18 Weeks
  Measured by changes in the modified Godin leisure questionnaire survey scores. The more minutes per week spent in exercise the better the physical activity.
Physical activity | From Baseline to 18 Weeks
  Measured by Fitbit data changes. The higher the step count the better the physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jethro Hu, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Pacific Neuroscience Institute / Saint John's Cancer Institute, Santa Monica, California
  - Duke University, Durham, North Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No